CLINICAL TRIAL: NCT06255509
Title: Dengue Virus Infection Amongst Patients With Acute Febrile Illness: Clinical Characteristics, Molecular and Serological Profiles for Vaccine Trial and Roll-out
Brief Title: Dengue Virus Infection Amongst Patients With Acute Febrile Illness
Status: Recruiting | Type: Observational
Sponsor: Tangerang District Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 445/068/KEP-RSUTNG
Record Dates: First submitted 2024-01-18; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Dengue
Keywords: Acute febrile illness; Dengue; Serotype
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational study that will be conducted in Tangerang Regency, Indonesia with primary objective to determine the clinical characteristics, specific immune responses, and viral serotypes in patients with confirmed dengue virus infection in Tangerang District, Indonesia.

DETAILED DESCRIPTION:
Dengue is a significant public health problem in Indonesia, with reported cases varies between 25.000-79.000 each year in 2013-2022. The disease is caused by four serotypes of Dengue virus (DENV-1, DENV-2, DENV-3, and DENV-4), transmitted primarily by the Aedes aegypti. However, dengue infection of DEN-4 are rarely reported compared to other dengue serotypes, such as in Vietnam, Philippines, and other Asian or other Latin American countries.

In Indonesia, DEN-4 was also the least serotypes reported. In contrast, DEN-4 is often found during dengue outbreaks. This findings has been reported in Jakarta and Jember outbreaks reports. The low prevalence of DEN-4 maybe because most studies was conducted in hospitals. Also, NS-1 RDT that is used for test has low sensitivity for DEN-4, particularly in secondary infection.

Overcoming the limitation the current diagnostic methods is critical for quick and precise treatment for individuals with dengue infection. Particularly, in the context for vaccine development and clinical trial. We chose Tangerang because it has a high risk of dengue virus transmission due to it is heavily populated area. Dengue remain a significant health problem as 50-100 cases reported each year from Public Health Centers, and >200 patients were hospitalized due to Dengue infection.

Therefore, this study will be conducted at 2 Public Health Centers (Kelapa Dua and Bojong Nangka) and Tangerang District Hospital for 1 year starting from 2 February 2024 to 31 January 2025.

Patient will be recruited when they satisfy inclusion and exclusion criteria and will be tested for RDT test and hematologic test. Blood and clinical data will be obtained from enrolled participant on enrollment and maximum 2 weeks after enrollment. Acute specimens from enrollment will be tested for NS1, IgM/ IgG using ELISA and molecular by PRNT while the convalescent specimen will be tested for IgG and IgM only. A subset of positive cases by PCR will be cultured and tested for PRNT.

Acute specimen from undiagnosed dengue infection will be tested for other pathogens.

Clinical and laboratory data will be analyzed for proportion for dengue among acute fever, proportion for each dengue serotypes, and clinical manifestation for each serotypes will be compared for severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 4 years old with fever (≥ 37.5°C), history of fever with antipyretic use, lasting less than or equal to 7 days
* Presence at least one of the following dengue-like symptoms:

  * Headache
  * Retro-orbital pain
  * Nausea/ vomiting
  * Muscle, bone, or joint pain
  * Rash or bleeding manifestations
* Patient or patient's guardian giving consent to participate in the study

Exclusion Criteria:

* Have a condition that may interfere with study procedures and compliance (based on doctor's assessment)
* Suspected of focal infection

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200 hospitalized patients and 200 public health center whom fulfill inclusion criteria and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2025-02-04 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
clinical characteristics | 1 year
  fever (yes/no), headache (yes/no), retro-orbital pain(yes/no), nausea/ vomiting (yes/no), arthralgia/ myalgia (yes/no), bleeding manifestation (yes/no)
haematologic profile | 1 year
  leukosit absolute (number/ ul), platelet (number/ul)
Rapid test for dengue | 1 year
  NS1 (positive/negative), IgM (positive/negative), IgG (positive/negative)
molecular (PCR) | 1 year
  DEN-1 (positive/negative), DEN-2 (positive/negative), DEN-3 (positive/negative), DEN-4 (positive/negative)
PRNT | 1 year
  DEN-1 (titer), DEN-2 (titer), DEN-3 (titer), DEN-4 (titer)

SECONDARY OUTCOMES:
prevalence of dengue virus infection among patients with acute fever | 1 year
  prevalence of DEN-1, DEN-2, DEN-3, DEN-4 among patients with acute fever

CONTACTS AND LOCATIONS:
Locations (1):
- Tangerang District Hospital, Tangerang, Banten, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT06255509/Prot_SAP_000.pdf